CLINICAL TRIAL: NCT00959088
Title: Faster AFB Identification, Speciation of TB, and Evaluation of Drug Resistance in HIV-Infected Persons Initiating TB Treatment
Brief Title: Faster Identification of TB and Evaluation of Drug Resistance in HIV-infected People
Acronym: FASTER
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5255; 1U01AI068636 (NIH); FASTER
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — samples of sputum and blood may be retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: HIV-infected individuals with suspected TB co-infection.

SUMMARY:
Early identification of tuberculosis (TB) is of particular importance in HIV-infected individuals, as a delay of therapy can be devastating in those with compromised immune systems. Diagnosis of TB in HIV is difficult, however, because 24-61% of HIV co-infected individuals with pulmonary TB have negative TB test results. In addition, conventional testing can take 6 weeks or longer and may not be available at all in many settings. This study is being conducted to see whether some new tests for identifying TB and for identifying resistance to TB drugs are at least as accurate as the current testing methods when used on HIV-infected individuals. The study will also assess whether the new tests can provide accurate results faster than the current methods.

DETAILED DESCRIPTION:
Early diagnosis of tuberculosis (TB) is of particular importance in HIV-infected individuals, as a delay of therapy can be devastating in those with compromised immune systems. Diagnosis of TB in HIV can be a particular challenge, however, because 24-61% of HIV co-infected individuals with pulmonary TB are smear-negative. Conventional solid media-based culture can take 6 weeks or longer for mycobacterial growth, and may not be available at all in many settings. The purpose of this study is to determine whether new tests for identifying TB and resistance to TB drugs are as effective as current tests and if these new tests can provide accurate results faster than the current method of testing for TB and drug resistance.

This trial will enroll HIV-infected individuals who are suspected to be co-infected with TB. Participants may be in this trial for up to nine months, depending on their test results. During the study, participants will provide one or two sputum samples, have a chest x-ray, and may have blood collected.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented at any time prior to study entry by a rapid HIV test or any licensed ELISA test kit
* Probable or confirmed pulmonary TB at the time of enrollment
* Current use of an anti-TB regimen for treatment of active TB for fewer than 7 days prior to sputum sample collection or anticipated initiation of same within 30 days after study entry
* Ability and willingness of participant or legal guardian/representative to provide informed consent.

Exclusion Criteria

* Receipt of 7 or more cumulative days of anti-TB treatment within 12 months prior to sputum collection
* Inability to provide sputum sample

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected individuals with suspected TB co-infection
Sampling Method: Non-Probability Sample
Enrollment: 641 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
GenoType Direct line probe assay result (MTB-positive or negative) and conventional mycobacterial culture assay result (MTB-positive or negative) on direct sputum samples | Throughout study

SECONDARY OUTCOMES:
GenoType Direct line probe assay results on direct sputum samples | Throughout study
GenoType MTBDR Plus line probe assay results on cultured and direct sputum samples | Throughout study
Identified strains of drug resistant MTB | Throughout study
AFB smear with ZN staining results | Throughout study
AFB smear as evaluated with fluorescent microscopy results | Throughout study
MTB culture results (including speciation and, if indicated, drug susceptibility) | Throughout study
MTB blood culture results | Throughout study
Follow up clinical assessment of MTB disease status | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Annie Luetkemeyer, MD, Study Chair — San Francisco General Hospital; Cynthia (Cindy) Firnhaber, MD, Study Chair — University of Witwatersrand, South Africa
Locations (3):
- Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro, Brazil
- Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima, Peru
- Wits HIV CRS, Johannesburg, Gauteng, South Africa